CLINICAL TRIAL: NCT00709176
Title: Outcomes of Triaged Family Care in Advanced Cancer
Acronym: FOCUS-Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Laurel L. Northouse, Ph.D. / Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01CA107383 (NIH); R01CA107383 (NIH); UMCC 2003-094 (Other: University of Michigan); IRBMED No. 2004-0129 (Other: University of Michigan)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Cancer
Keywords: Quality of Life; Randomized Clinical Trial; Advanced Cancer; Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Family caregiver; cancer survivorship; coping; communication; uncertainty; support; depression; self-efficacy; benefits of illness; Caregivers
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Communication; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief (Experimental): Dyads randomized to BRIEF arm received the Brief FOCUS Program (two home visits and one phone call by a trained nurse) in addition to standard clinical care.
  Interventions: Behavioral: Brief FOCUS Program
- Extensive (Experimental): Dyads randomized to EXTENSIVE arm received the Extensive FOCUS Program (4 home visits and two phone calls by a trained nurse) in addition to standard clinical care.
  Interventions: Behavioral: Extensive FOCUS Program
- Control (No Intervention): Dyads randomized to CONTROL arm continued with standard clinical care.

INTERVENTIONS:
Behavioral: Brief FOCUS Program — Dyads randomized to this arm received the FOCUS Brief Program, two home visits and one phone call by a trained nurse.
  Other Names: Family(F),Optimism(O),Coping(C),Uncertainty(U),Symptoms(S); Family-based Intervention; Cancer Patient and Family Member Intervention
  Arms: Brief
Behavioral: Extensive FOCUS Program — Dyads randomized to this arm received the FOCUS Extensive Program, 4 home visits and two phone calls by a trained nurse.
  Other Names: Family(F),Optimism(O),Coping(C),Uncertainty(U),Symptoms(S); Family-based Intervention; Cancer Patient and Family Member Intervention
  Arms: Extensive

SUMMARY:
The purpose of this study is to assess the quality of life of patients with advanced cancer and their family caregivers and to evaluate two doses of a family-based program of care versus control.

DETAILED DESCRIPTION:
The purpose of this study is to:

1. determine if family dyads randomly assigned to either a brief or extensive family-based program of care have better proximal and distal outcomes from both a clinical and economic perspective than dyads randomly assigned to usual care
2. determine if the brief or extensive program of care has a differential effect on patient and caregiver outcomes depending on the patient's baseline risk for distress status (high versus low).

A longitudinal, randomized clinical trial is being used for patients with advanced lung, colorectal, prostate, and breast cancer and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage 3 or 4 breast, prostate, colorectal and lung cancers.
* Patients must be 21 years old or older, physically and mentally able to participate, speak and understand English, have a minimum life expectancy of six months, live within 75 miles of one of the participating sites and have a family caregiver who is willing to participate in the study.
* For this study "family caregiver" is defined as the person who provides the patient with physical and/or emotional support during cancer treatment.
* Family caregivers must be 18 years old or older, physically and mentally able to participate, and speak and understand English.

Exclusion Criteria:

* Patients will be excluded if they have multiple primary cancer sites.
* Family caregivers will be excluded if they, themselves, have been diagnosed with cancer during the previous year and/or are in active treatment for cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, 3 and 6 months

SECONDARY OUTCOMES:
Risk for Distress | Baseline
Change in Emotional Distress | Baseline, 3 and 6 months
Change in Appraisal of Illness/Caregiving | Baseline, 3 and 6 months
Change in Uncertainty | Baseline, 3 and 6 months
Change in Hopelessness | Baseline, 3 and 6 months
Change in Self-efficacy | Baseline, 3 and 6 months
Change in Benefits of Illness | Baseline, 3 and 6 months
Change in Family Communication | Baseline, 3 and 6 months
Change in Support | Baseline, 3 and 6 months
Change in Depression | Baseline, 3 and 6 months
Change in Coping | Baseline, 3 and 6 months
Change in Health Care Resource Utilization | Baseline, 3 and 6 months
Change in Caregiver Burden | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurel L Northouse, PhD, RN, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - St. Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Providence Hospital Cancer Institute, Southfield, Michigan

REFERENCES:
- [Background] Northouse L. Helping families of patients with cancer. Oncol Nurs Forum. 2005 Jul 1;32(4):743-50. doi: 10.1188/05.onf.743-750. PMID 15990903
- [Result] Northouse LL, Mood DW, Schafenacker A, Kalemkerian G, Zalupski M, LoRusso P, Hayes DF, Hussain M, Ruckdeschel J, Fendrick AM, Trask PC, Ronis DL, Kershaw T. Randomized clinical trial of a brief and extensive dyadic intervention for advanced cancer patients and their family caregivers. Psychooncology. 2013 Mar;22(3):555-63. doi: 10.1002/pon.3036. Epub 2012 Jan 31. PMID 22290823
- [Derived] Guan T, Chapman MV, de Saxe Zerden L, Zimmer C, Braden CJ, Rizo CF, Northouse L, Song L. Illness uncertainty and quality of life in patients with advanced cancer and their family caregivers: An actor-partner interdependence model analysis. Psychooncology. 2023 Nov;32(11):1744-1751. doi: 10.1002/pon.6228. Epub 2023 Oct 4. PMID 37794604
- See also: University of Michigan Comprehensive Cancer Center website — http://www.cancer.med.umich.edu/